CLINICAL TRIAL: NCT03666975
Title: Investigating Vibration Therapy on Rate of Growth in Length of Shorter Leg of Children 6-12 Years With Leg-length Discrepancy (LLD): a Pilot Randomised Trial of Different Low Intensity Vibration (LIV) Therapy.
Brief Title: Can we Promote Bone Lengthening With Vibration Therapy?
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Principal Investigator, Mary Fewtrell, Professor of Paediatric Nutrition, University College, London
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 210984
Record Dates: First submitted 2018-08-23; First posted 2018-09-12 (Actual); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Leg Length Discrepancy; Leg Length Difference
Keywords: Low intensity vibration; Paediatric bone growth
MeSH Terms: conditions — Leg Length Inequality

STUDY DESIGN:
Intervention Model Description: Vibration therapy intervention study involving children with pre-existing LLD to be assessed monthly for 4 months and then randomised to have one of 2 vibration therapies for three months and finally 6 months leg-length measurements to assess changes in extra bone length achieved in the shorter leg during the intervention.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Blinding / masking of participants investigator and assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- LIV 30 Hz, 0.4 g (Experimental): LIV 30 Hz, 0.4 g Low intensity vibration to short leg 3x / week x 10 wks
  Interventions: Device: LIV 30 Hz
- LIV 30 Hz, 1.0 g (Experimental): LIV 30 Hz, 1.0 g Low intensity vibration to short leg 3x/week x 10 wks
  Interventions: Device: LIV 30 Hz

INTERVENTIONS:
Device: LIV 30 Hz — LivMD LIV platform
  Other Names: Low intensity vibration medical device (LivMD) platform

SUMMARY:
This research will assess whether vibration therapy can increase bone-growth in length of the shorter leg in children aged 6-12 years with pre-existing leg length difference (LLD) which is being treated with a heel-raise or orthotics. Children will be referred by orthopaedic and musculoskeletal clinics, physiotherapists and orthotists. Children will have monthly measurement of leg length (LL) over a 13 month period (4 months pre-treatment, 3 months treatment, 6 months post-treatment) using a portable Ultrasound-laser system which is safe, accurate, reproducible and validated against standing x-ray measurement. During the treatment phase they will be randomised to receive vibration therapy 3 times per week using a vibration platform at 30 Hz and very low amplitude of 0.4g (less than experienced when walking) or 30 Hz at 1.0 g (the same force as standing with the effect of gravity). The child will stand with the shorter leg on the platform and the longer leg on a stationary block for 15 minutes per treatment session. The aim is to assess the potential of this safe, non-invasive and potentially cost-effective method for levelling LL. If effective, the research could be extended in future to children with much larger LLD in whom it could potentially avoid the need for surgery and minimise long-term musculoskeletal disability.

DETAILED DESCRIPTION:
Subjects with a documented treatment history for LLD will be recruited via orthopaedic, orthotic, physiotherapy and musculoskeletal clinical practitioners in London.

All specialist practitioners and clinics across London will be informed about the study (via Practitioner/LLD Letter), asking them to forward information direct to eligible subjects .

20-25 subjects with pre-existing LLD who are undergoing treatment with shoe raises, heel-lifts or built-up shoes will be recruited. Parents receiving the Parental information sheet outlining the study are therein invited to contact the researchers who will arrange a baseline visit to the clinic. At this visit, the study will be discussed and all questions answered. If the child and family are willing to take part, written informed consent will be taken from the parent and assent from the child. Baseline measurements will be taken as below.

Treatment of subjects:

All subjects will have accurate LL measurement at baseline and then LL measurement monthly over 13 months (4 months pre-treatment, 3 months intervention and 6 months follow-up).

Subjects at the 4th month will start intervention with LIV and will attend the clinic 3 times per week. Some subjects living further away will use a loaned LIV platform at home for treatment and will be trained in its correct use. They will be asked to send in weekly reports of the number of sessions and minutes per session on the platform. The research team will keep an accurate note of total time. Subjects who have a machine at home will be asked to use the treatment at least 3 times per week, but that they can use it once per day if they wish; they will be asked to record the exact time spent on the platform. All monthly leg-length measurements will take place at the study clinic at a time to suit the family.

All subjects will use the following low intensity vibration intervention: 0.4 g and 30 Hz based on the fact that this is the 'low intensity vibration medical device' (LIVMD) machine, developed by Professor Clinton Rubin for use by NASA astronauts that conforms to all IS0 safety measures.

The primary outcome measure will be the difference in LL growth of the treated vs. untreated leg over the intervention period. Height and weight of all subjects will be taken monthly and their level of physical activity (0-5) and any high-performance sports activity such as trampoline or plyometrics training (on a scale of 0-5) will be assessed by questionnaire. Previous lower limb dysfunction, injury, fracture or surgery, ongoing illness, drug treatment, growth hormone treatment or use of shoe heel-raise will also be assessed by questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* age 6-12 years
* pre-existing leg length difference (LLD) currently being treated by a practitioner with heel raise or orthotics

Exclusion Criteria:

* history of Osteogenesis Imperfecta (OI) or bone growth dysfunction
* history of lower limb deformities, fractures or surgery.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2017-01-28 (Actual); Primary Completion 2018-12-28 (Estimated); Study Completion 2018-12-28 (Estimated)

PRIMARY OUTCOMES:
Difference between treatment groups in LL growth of the treated v untreated leg over the intervention period. | 3 months
  LASER and ultrasound measurements of both legs will be taken monthly during the treatment (months 4-7) phase (unit mm).

SECONDARY OUTCOMES:
Difference in growth of the treated and untreated leg within each subject over the pre-treatment (4 months) and post-treatment (6 months) periods. | 10 months
  LL measurements as for primary outcome - in mm 2. Within-subject differences in growth between treated and untreated legs, compared at pre-treatment and treatment phases. Unit of measurement = mm

CONTACTS AND LOCATIONS:
Overall Officials: Mary Fewtrell, Principal Investigator — UCL London
Locations (1):
- Gosh Ich-Ucl, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No